CLINICAL TRIAL: NCT04437524
Title: Comparison of the Effects of Balance-proprioception and Aerobic Exercises on Functional Status, Pain and Strength Parameters in Patients With Fibromyalgia Syndrome (FMS).
Brief Title: Comparison of the Effects of Balance-proprioception and Aerobic Exercises on Functional Status and Strength Parameters in Patients With Fibromyalgia.
Acronym: FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Hadi Yavuz, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 196481654
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia, aerobic exercise, balance, proprioception, pain, strength
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balance-proprioception exercises group (Active Comparator): balance-proprioception exercises group
  Interventions: Other: therapeutic exercises
- aerobic exercises group (Active Comparator): aerobic exercises group
  Interventions: Other: therapeutic exercises

INTERVENTIONS:
Other: therapeutic exercises — Treatment that will continue 3 days a week for 6 weeks in female patients with fibromyalgia.

SUMMARY:
In this study, it was aimed to examine the effects of aerobic exercise and balance-proprioception exercises on pain, functionality and strength parameters of fibromyalgia patients and to compare the two exercise types.

DETAILED DESCRIPTION:
In the study planned to evaluate the effect of aerobic and balance-proprioception exercises on the symptoms of the disease and the superiority of the two exercise models in patients with fibromyalgia syndrom (FMS), 62 women who meet the inclusion criteria will be randomly divided into two groups. Aerobic exercise group (n = 26) and balance-proprioception exercise group (n = 26) will be applied for 3 weeks a week, 6 days a week under the supervision of a physiotherapist in the exercise laboratory of the Istanbul Medical Faculty Sports Medicine Department. Pain (VAS), functional status (FİQ) and knee extension muscle strength (Cybex isokinetic dynamometer) will be evaluated before and after the program. Cognitive status will be evaluated with standardized Mini Mental Test only before the program.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 60,
* Symptoms lasting longer than 3 months,
* According to the 2013 ACR criteria, the Pain Settlement Score (PLI) is ≥17,
* According to the 2013 ACR criteria, the Symptomatic Impact Scoring (SIQR) is ≥21,
* Acceptance of treatment that will continue 3 days a week for 6 weeks,
* The possibility of any change in medical treatment due to FMS during the study is not foreseen.

Exclusion Criteria:

* Known central or peripheral nervous system disease, progressive neurological damage,
* Any serious cardiovascular pathology,
* Sense, loss of sense of position, unhealed fracture or a surgical wound,
* Presence of uncontrolled hypertension,
* Failure to understand or perform simple commands.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female fibromyalgia patients will be admitted to the study.
Enrollment: 51 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 6 weeks
  In order to evaluate the functional status in patients with FMS, FIQ Burchardt et al. It is a specific scale developed by. FIQ consists of 10 items. Calculation is made so that the upper limit of each item is 10 points. The maximum score that can be reached is 100. A high total score indicates that the person is more affected by the disease.
Pain (Visual Analogue Scale) | 6 weeks
  Visual Analaog Scale is used to measure the severity of pain in patients. The patient is told that there is no "0" pain on the 10 cm ruler drawn on paper, "10" is the most experienced pain, and the patient is asked to mark on the ruler according to the severity of the pain he/she feels. The distance of the marked point from zero is recorded as the Visual Analogue Scale score in cm.
Muscle Strength Evaluation | 6 weeks
  The CSMI Humac Norm 2015 isokinetic dynamometer will be used to evaluate muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Metin, Professor, Study Director — İstanbul Univesity, İstanbul Faculty of Medicine
Locations (1):
- İstanbul Faculty of Medicine, Department of Sports Medicine, Istanbul, Turkey (Türkiye)